CLINICAL TRIAL: NCT00834704
Title: Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, Pharmacodynamic, and Pharmacokinetic Study of PEGPH20 (PEGylated Recombinant Human Hyaluronidase) Given Intravenously to Patients With Advanced Solid Tumors
Brief Title: Safety Study of PEGPH20 Given to Patients With Advanced Solid Tumors
Acronym: PEG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HALO-109-101
Record Dates: First submitted 2009-01-29; First posted 2009-02-03 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2012-09

CONDITIONS: Solid Tumor
Keywords: PEGPH20; PEGylated recombinant human hyaluronidase; Metastatic or locally advanced solid tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — PEGPH20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Dose determination
  Interventions: Drug: PEGPH20

INTERVENTIONS:
Drug: PEGPH20 — PEGylated recombinant human hyaluronidase

SUMMARY:
Open-label, multicenter, dose-escalation, safety, pharmacodynamic, and pharmacokinetic study.

DETAILED DESCRIPTION:
This is a study of PEGPH20 in human subjects and is designed to evaluate the safety of PEGPH20 and to determine the maximum tolerated dose of PEGPH20. All patients will receive PEGPH20. Each group of patients will receive a higher dose than the previous group. This will continue until the group with the highest planned dose completes the study or until a group has major side effects from their assigned dose.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic (histologic or cytologic) confirmation of metastatic or locally advanced solid tumor.
* Patients who have experienced disease progression after receiving appropriate standard / approved chemotherapy and for whom no further standard or palliative treatment measures exist, or who have chosen to decline standard or palliative treatment.
* One or more tumors measurable by RECIST criteria.
* Karnofsky performance status ≥ 70%.
* Recovery from any toxic or other effects of all previous therapy, including radiation, chemotherapy and surgery.
* Negative serum or urine pregnancy test result in women of childbearing potential.
* For men and women of child-producing potential, agreement to use effective contraception (hormonal or barrier birth control or abstinence) from the time of screening before study entry and throughout study participation.

Exclusion Criteria:

* Brain metastasis.
* New York Heart Association Class III or IV cardiac disease, myocardial infarction, or cardiac arrhythmia requiring medical therapy.
* Known allergy to hyaluronidase.
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions including psychiatric illness) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* Women currently breast feeding.
* Concurrent participation in any other interventional therapeutic study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine the recommended phase 2 dose (RP2D) of PEGPH20. To evaluate the safety and tolerability of PEGPH20 in advanced cancer patients over a range of doses. | 28 days

SECONDARY OUTCOMES:
To determine the pharmacokinetics (PK) of PEGPH20 | 28 days
To determine the dose-limiting toxicities (DLTs) of PEGPH20. | 28 days
To observe patients for any evidence of anti-tumor activity (efficacy). | 28 days
To explore pharmacodynamic endpoints that may guide the further development of PEGPH20. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Joy Zhu, M.D., Study Director — Halozyme Therapeutics
Locations (3):
- United States (3):
  - T Gen Clinical Research Services, Scottsdale, Arizona
  - Premiere Oncology, Santa Monica, California
  - Sarah Cannon Research Institute, Nashville, Tennessee